CLINICAL TRIAL: NCT01038180
Title: Complications Following Pacemaker or ICD Implantation: Results From The Danish Pacemaker and ICD Register
Brief Title: Complications Following Pacemaker Implantation
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Rikke Esberg Kirkfeldt, Aarhus Universityhospital, Skejby
Other Study IDs: SKS-REK-1
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Bradycardia
Keywords: pacemaker; adverse effects
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pacemaker group

SUMMARY:
This study examines possible risk factors with regard to complications following pacemaker implantation.

DETAILED DESCRIPTION:
This study examines possible risk factors with regard to complications following pacemaker implantation. We are using data from The Danish Pacemaker Register.

ELIGIBILITY:
Inclusion Criteria:

* permanent cardiac pacemaker

Exclusion Criteria:none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Danish patients receiving a permanent cardiac pacemaker during the years 1997 to 2008
Sampling Method: Probability Sample
Enrollment: 28000 (Actual)
Dates: Start 1997-01; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rikke E Kirkfeldt, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Kirkfeldt RE, Johansen JB, Nohr EA, Moller M, Arnsbo P, Nielsen JC. Risk factors for lead complications in cardiac pacing: a population-based cohort study of 28,860 Danish patients. Heart Rhythm. 2011 Oct;8(10):1622-8. doi: 10.1016/j.hrthm.2011.04.014. Epub 2011 Apr 14. PMID 21699827